CLINICAL TRIAL: NCT03004664
Title: A Patient-Centered Framework to Test the Comparative Effectiveness of Culturally and Contextually Appropriate Program Options for Latinos With Diabetes From Low-Income Households
Brief Title: Comparing Program Options for Latinos With Diabetes
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Janet M Page-Reeves, Research Assistant Professor, University of New Mexico
Other Study IDs: 16-303
Record Dates: First submitted 2016-12-16; First posted 2016-12-29 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus
Keywords: Latinos; Low Income; Self Management; Education; Cultural Competence
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Support Empowerment Model: The Center for Diabetes Education at the University of New Mexico Hospital (CDE) uses the Diabetes Self-Management Support Empowerment Model (DSMS). The DSMS combines a series of clinically informed group didactic sessions that use a patient self-determination approach to empower patients to take control of their own diabetes health with follow-up supports to sustain self-management gains achieved during the sessions. Patients attend a six-week group instructional session with 9 hours of class plus an individual follow-up with a certified diabetes educator. The group sessions have discussion supported by didactic conversation "maps" where the facilitator guides but does not control the conversation based on session thematic goals.
  Interventions: Behavioral: Support Empowerment Model
- The Chronic Care Model: One Hope Centro de Vida Diabetes Program is based on the Chronic Care Model (CCM). The CCM involves 6 synergistic domains: 1.) Improved access to care, 2.) Patient self-management support, 3.) Patient decision support, 4.) Care coordination, 5.) Integrated health information systems, and 6.) Access to community resources. To create a holistic care regime, the CCM focuses on addressing social determinants of health by meeting the medical, cultural, and linguistic needs of patients through integration of cultural norms and social relationships from the patient population into program design.
  Interventions: Behavioral: The Chronic Care Model

INTERVENTIONS:
Behavioral: Support Empowerment Model — The DSMS combines a series of clinically informed group didactic sessions that use a patient self-determination approach to empower patients to take control of their own diabetes health with follow-up supports to sustain self-management gains achieved during the sessions.
  Other Names: Diabetes Self-Management Support Empowerment Model
  Groups: Support Empowerment Model
Behavioral: The Chronic Care Model — the CCM focuses on addressing social determinants of health by meeting the medical, cultural, and linguistic needs of patients through integration of cultural norms and social relationships from the patient population into program design
  Groups: The Chronic Care Model

SUMMARY:
BACKGROUND AND SIGNIFICANCE:

Diabetes is a national health problem, yet Latinos from low-income households are at greater risk. Although guidelines recommend that patients learn self-management strategies, many people are not able to do so effectively and cannot control their diabetes. Studies show that culturally competent self-management programming can help, but patients in preliminary research indicated that not all programs sufficiently respect patients' cultural values or account for their socio-economic limitations.

STUDY AIMS:

This project will compare two models for culturally competent diabetes self-management programming. The hypothesis is that the program model that best considers patient culture and accommodates patient socio-economic circumstances will have the best outcomes.

COMPARATORS:

2 diabetes self-management program models used by many Latino patients from low-income households in Albuquerque, New Mexico

1. The Diabetes Self-Management Support Empowerment Model
2. The Chronic Care Model

STUDY POPULATION:

Patients will be 240 individuals who consider themselves to be Latino and who are from low-income households. In addition, 240 patients will identify a corresponding social support to participate with them. Outcomes will be measured based on the 240 patient participants. Social support data will be measured as a covariate to understand patient outcomes.

PRIMARY OUTCOME:

Improved capacity for diabetes self-management measured as diabetes knowledge and patient activation or the ability to put that knowledge into action.

SECONDARY OUTCOME:

Successful diabetes self-management measured through reduced A1c, BMI and depression. Patient stress levels will also be measured using testing of hair samples to identify levels of cortisol as a biological marker for chronic stress.

METHODS:

Statistical calculations will be conducted to make sure that the things being compared are differences in program design and not differences in individual patient characteristics. This study will compare whether the programs improve diabetes health knowledge, ability to act, and A1c, BMI, depression and stress control, and determine which program is the best.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE:

Diabetes is a national health priority but diabetes risk is extremely high for Latinos from low-income households. Health guidelines recommend that individuals learn strategies to self-management their diabetes, but getting people to adopt required lifestyle changes is challenging and many people are not able to prevent their pre-diabetes from escalating or to control their diabetes. Systematic reviews show that culturally competent self-management programming can significantly improve diabetes outcomes, and different models for culturally competent programming have been developed.

STUDY AIMS:

The goal of this study is to compare the effectiveness of 2 distinct evidence-based models for culturally competent diabetes health promotion. The hypothesis is that the program model that interfaces most synergistically with patient's culture and everyday life circumstances will have the best diabetes health outcomes.

Aim 1: Characterize the ways that three culturally competent diabetes self-management programs interface with patient culture and socioeconomic context

Aim 2: Measure and compare improvement in patient capacity for diabetes self-management.

Aim 3: Measure and compare patient success at self-management Study Description

OVERALL STUDY DESIGN:

This study follows NIH standards for mixed-method research by integrating data from quantitative and qualitative components of the study in an iterative fashion. The sample size and power estimates are based on realistic evaluation of effect size. Data collection will involve programmatic assessments, interviews, focus groups, surveys, and testing for A1c, BMI, and stress. The research team has the expertise and experience in patient-engaged research necessary to conduct the proposed study and the investigators have an institutional infrastructure that supports the academic and community partnerships necessary for this study.

MAIN COMPONENTS OF THE INTERVENTION AND COMPARATORS:

This study compares 2 diabetes self-management programs that serve a large Latino patient population from low-income households in Albuquerque, New Mexico

1. The Diabetes Self-Management Support Empowerment Model
2. The Chronic Care Model

PRIMARY & SECONDARY OUTCOMES:

PRIMARY: Improved capacity for diabetes self-management measured through improvements in diabetes knowledge and diabetes-related patient activation.

SECONDARY: Successful diabetes self-management.

ANALYTIC METHODS:

Descriptive statistics will be calculated to summarize patient characteristics. Means and standard deviations or medians and quartiles will be calculated for continuous variables and will be compared across site by ANOVA or Kruskal-Wallis test, depending on the distribution of the data. Frequencies and percentages will be calculated for categorical variables and will be compared with the chi-square test or Fisher's exact test, as appropriate. Significant differences will be noted and to adjust for possible confounding, those variables will be considered for inclusion as covariates in the analyses for the primary and secondary outcomes in addition to other clinically meaningful variables and their interactions. It is expected that patient characteristics to be similar across the two treatment sites; however, to control for potential differences in the populations, the investigators will adjust for potential confounding covariates by using propensity scores to stratify subjects into groups based on the probability that they attended a particular treatment site given particular demographic characteristics including sex, age, primary language, level of education, nativity, and type of insurance. Patients will be grouped by quintile of propensity score for a total of five strata and each will be analyzed for the primary and secondary outcomes independently. Analyses will be performed in standard statistical software. Propensity score matching allows for causal inference in our non-experimental settings by selecting similar subsets of comparison units between treatment groups across a high-dimensional set of pretreatment characteristics. For qualitative data, the investigators will conduct a rigorous, disciplined, empirical analysis based on plausibility, credibility and relevance. The investigators will conduct a theory-driven qualitative content analysis, reading through transcripts to identify conceptual categories and patterns related to specified domains of inquiry, creating a qualitative codebook, and developing conceptual summaries for each transcript. Following review and summary, the investigators will code transcripts for systematic themes and subthemes and explore interconnections between theme categories and develop a holistic interpretation of the data ("constant comparison").

ELIGIBILITY:
INCLUSION CRITERIA:

Patient Participants:

1. Adults (men and women) who have been identified by a provider as having pre-diabetes (A1c 5.7-6.4) or diabetes (A1c 6.5 or above)
2. Enter one of the two diabetes programs during the study
3. Self-identify as "Latino"
4. Can identify a social support or key member of their social network who will agree to participate with them
5. Are not pregnant (participants who become pregnant during the study will be excluded)
6. Have household income 250% of the Federal Poverty Level (FPL) or below.

Social support participants:

1. Adults
2. Individuals who are identified by the patient participants as their social support

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* Pregnant women

Participants who become pregnant during the study will be excluded. At enrollment and before each data collection appointment, female patient participants will be screened to specifically exclude those who are pregnant. There is no risk to a pregnant woman or a fetus entailed in participation in this study because the study only involves data collection from individuals who have been instructed to participate in a diabetes self-management program by their provider. However, pregnant individuals will be excluded because pregnancy could impact outcomes in a way that will influence scientific analysis of diabetes self-management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STUDY POPULATION:
  Patients will be identified through the diabetes programs at 2 sites: a total of 240 patient-caregiver pairs will be recruited: patients and a corresponding caregiver of each patient.
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Patients will improve their capacity for diabetes self-management: Measured through change in Diabetes Knowledge | (baseline to 3 months), (3 months to 6 months), (6 months to 12 months)
  Improvement in diabetes knowledge measured through change in scores on The Diabetes Knowledge Questionnaire [DKQ])
Patients will improve their capacity for diabetes self-management: Measured through change in Patient Activation | (baseline to 3 months), (3 months to 6 months), (6 months to 12 months)
  Improvement in patient ability to manage their own diabetes measured through changes in score on the Patient Activation Measure (PAM)

SECONDARY OUTCOMES:
Patients will successfully self-manage their diabetes measured through change (reduction) in their blood glucose | (baseline to 3 months), (3 months to 6 months), (6 months to 12 months)
  Reduction in their blood glucose as indicated by A1c 21
Patients will successfully self-manage their diabetes measured through change (reduction) in Body Mass Index (BMI) | (baseline to 3 months), (3 months to 6 months), (6 months to 12 months)
  Reduction in BMI
Patients will successfully self-manage their diabetes as measured through change (reduction) in depression | (baseline to 3 months), (3 months to 6 months), (6 months to 12 months)
  Reduction in depression measured through changes in depression index score in score on Patient Health Questionaire 9-Item set [PHQ-9])
Patients will successfully self-manage their diabetes as measured though change (reduction) in chronic stress levels | (baseline to 6 months), (6 months to 12 months)
  Improvement in chronic stress levels indicated through testing of hair sample for change (reduction) in circulating level of cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Page-Reeves, Ph.D., Principal Investigator — University of New Mexico School of Medicine
Locations (2):
- United States (2):
  - One Hope Centro de Vida Health Center, Albuquerque, New Mexico
  - University of New Mexico Hospital, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Page-Reeves J, Regino L, Murray-Krezan C, Bleecker M, Erhardt E, Burge M, Bearer E, Mishra S. A comparative effectiveness study of two culturally competent models of diabetes self-management programming for Latinos from low-income households. BMC Endocr Disord. 2017 Jul 24;17(1):46. doi: 10.1186/s12902-017-0192-4. PMID 28738902

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT03004664/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03004664/ICF_001.pdf